CLINICAL TRIAL: NCT06850038
Title: Prospective Registry-Based Study Evaluating the Effectiveness and Safety of Odevixibat in Participants With Alagille Syndrome (ALGS)
Brief Title: A Study Observing the Long-term, Effectiveness and Safety of Odevixibat (Bylvay) in Patients With Alagille Syndrome (ALGS) Who Are Receiving Ongoing Treatment
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60240-033
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will collect information from patients with Alagille syndrome (ALGS) as they use odevixibat (Bylvay) in their daily lives.

Odevixibat is a medicine that helps patients with ALGS, a rare disease that harms their liver and causes itching.

The main aim of this study is to observe the long-term, everyday effectiveness and safety of the drug odevixibat in patients with ALGS who are receiving ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALGS.
* On (or starting) active odevixibat treatment.
* Signed informed consent and assent, as appropriate. Consent/assent from the participant or legal representative should be obtained, as appropriate, before any study data collection is conducted. Participants who turn 18 years of age (or legal age per country) while participating in the study will be required to provide consent for themselves.

Exclusion Criteria:

* Currently participating in a clinical trial with odevixibat.
* Currently participating in any interventional clinical trial for ALGS.
* Have any contraindication to odevixibat as per the locally approved label.
* Had liver transplant before enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with ALGS who start treatment with odevixibat (Bylvay) will be enrolled into the registry. Patients who started odevixibat treatment before the implementation of the registry study may also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Alagille syndrome (ALGS) who are treated with odevixibat and undergo biliary diversion surgery or liver transplantation. | From first dose to end of study (approximately 5 years data collection)
Surgical biliary diversion-free survival | From first dose to end of study (approximately 5 years data collection)
  Defined as time from the start of odevixibat treatment to the first occurrence of surgical biliary diversion or death.
Liver transplant-free survival | From first dose to end of study (approximately 5 years data collection)
  Defined as time from the start of odevixibat treatment to the first occurrence of liver transplant or death.
Overall survival | From first dose to end of study (approximately 5 years data collection)
  Defined as time from the start of odevixibat treatment to death.

SECONDARY OUTCOMES:
Change from Baseline in Weight | From first dose to end of study (approximately 5 years data collection)
  This endpoint will measure the change in participants' weight from baseline, reported as standard-deviation scores (z-scores) to account for age and sex-specific growth variations.
Change from Baseline in Height | From first dose to end of study (approximately 5 years data collection)
  This endpoint will measure the change in participants' height from baseline, reported as standard-deviation scores (z-scores) to account for age and sex-specific growth variations.
Percentage of participants with Adverse Events (AEs) associated with fat-soluble vitamin (FSV) deficiencies and their possible sequelae. | From signing of the Informed Consent Form (ICF) to 180 days after the last dose intake of odevixibat
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with suspected hepatotoxic Adverse events (AEs) requiring interruption of odevixibat | From signing of the ICF to 180 days after the last dose intake of odevixibat
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with bleeding AEs | From signing of the ICF to 180 days after the last dose intake of odevixibat
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with AEs | From signing of the ICF to 180 days after the last dose intake of odevixibat
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (3):
- United States (3):
  - NYU Langone - NYU Grossman School of Medicine, New York, New York
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Proactive El Paso,LLC, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/